CLINICAL TRIAL: NCT04940455
Title: Effect of Realistic Simulation and Digital Educational Platforms for Learning Nursing Student: Randomized Clinical Trial
Brief Title: Effect of Realistic Simulation and Digital Educational Platforms for Learning Nursing Student
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Brasilia (Other)
Responsible Party: Principal Investigator, Marcia Cristina da Silva Magro, Principal Investigador, PhD, University of Brasilia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 28233120.4.0000.0030
Record Dates: First submitted 2021-06-17; First posted 2021-06-25 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Educational Technology
Keywords: Educational Technology; Simulation Training; "Learning"; Learning Curve; Active Learning; Nursing

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational digital platforms (Experimental): Nursing students from the Experimental Group (GE), will participate in educational activities made available on digital platforms on "nursing care for patients with signs and symptoms of sepsis"
  Interventions: Other: Educational digital platforms
- High-Fidelity Simulation (Active Comparator): Nursing students in the Control Group (GC) will be exposed to high-fidelity simulation in the intensive care setting, where they must solve situations and procedures related to the nurse's performance in recognizing the signs and symptoms of sepsis.
  Interventions: Other: Educational digital platforms

INTERVENTIONS:
Other: Educational digital platforms — The digital educational platforms will be implemented through games of questions and answers, simulated cases sent via google forms about the nurse's performance in a critical care unit facing the patient with signs and symptoms of sepsis. The questions in the games will aim to develop clinical judgment and quick decision-making in nursing students in order not to compromise the health care of the patient in sepsis.

SUMMARY:
Teaching modalities that integrate digital educational technologies, such as educational games, dummies and simulated environments, develop critical thinking in students, the absorption of significant learning and the consequent reduction in the exposure of patients to the damage associated with health care. Thus, this study will evaluate the effectiveness of simulation strategies and digital educational platforms in the teaching-learning process, in self-confidence and its implications for the physiological variables and stressful feelings of undergraduate nursing students. Our hypothesis is that students submitted to the use of digital platforms will present lower levels of self-efficacy, capacity for clinical judgment and retention of knowledge when compared to those who were submitted to the simulation strategy.

DETAILED DESCRIPTION:
The study will be carried out in the simulation laboratory of two Higher Education Institutions, one public and the other private in the city of Brasília, Brazil. The sample will consist of 100 students randomized into an experimental group (n=50) and a control group (n=50). Students enrolled in the undergraduate nursing course, aged 18 years or over, will be eligible; have minimal approval in a discipline related to the content of "Nursing Care for Adult Patients". Students who work actively in the scenario of patient care in critical and risk situations will be excluded; members of the Academic League of Realistic Health Simulation and those with prior training in the health field. It is expected that nursing students, through active and innovative strategies, will be able to obtain and retain greater knowledge, raise levels of self-efficacy and clinical judgment, for their performance in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

Aged over 18 years;

Students approved in the discipline related to nursing care for adult and elderly patients.

Exclusion Criteria:

Students who actively work in the scenario of patient care in critical and risk situations; Members of the Realistic Health Simulation League; Students with previous training in the health area (nursing technicians, firefighters, among others) ; Participants who for some reason are absent from one of the project stages.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Cognitive Performance (Baseline) | Applied before the intervention
  Application of a questionnaire with ten multiple choice questions to assess the knowledge of nursing students about signs and sepsis symptoms
Cognitive Performance (Post-Test) | Applied immediately after the intervention
  Application of a questionnaire with ten multiple choice questions to assess the knowledge of nursing students about signs and sepsis symptoms
Cognitive Performance (Retention over time) | Applied thirty days after the intervention
  Application of a questionnaire with ten multiple choice questions to assess the knowledge of nursing students about signs and sepsis symptoms
Cognitive Performance (Retention over time) | Applied sixty days after the intervention
  Application of a questionnaire with ten multiple choice questions to assess the knowledge of nursing students about signs and sepsis symptoms
Clinical Judgment (Baseline) | Applied before the intervention
  Evaluation of the development of clinical reasoning of nursing students. The instrument Lasater clinical Judgment Rubric (LCJR)- Brazilian Version will be used. It assesses 11 dimensions at four levels of clinical judgment (recognition, interpretation, response, reflection). The total score ranges from 11 to 44, where the "initial" level generates one point, the "in development" level generates two points, the "proficient" level generates three points and the "exemplary" level generates four points.
Clinical Judgment | Applied immediately after the intervention
  Evaluation of the development of clinical reasoning of nursing students. The instrument Lasater clinical Judgment Rubric (LCJR) - Brazilian Version will be used. It assesses 11 dimensions at four levels of clinical judgment (recognition, interpretation, response, reflection). The total score ranges from 11 to 44, where the "initial" level generates one point, the "in development" level generates two points, the "proficient" level generates three points and the "exemplary" level generates four points .
Clinical Judgment | Applied thirty days after the intervention
  Evaluation of the development of clinical reasoning of nursing students. The instrument Lasater clinical Judgment Rubric (LCJR) - Brazilian Version will be used. It assesses 11 dimensions at four levels of clinical judgment (recognition, interpretation, response, reflection). The total score ranges from 11 to 44, where the "initial" level generates one point, the "in development" level generates two points, the "proficient" level generates three points and the "exemplary" level generates four points.
Clinical Judgment | Applied sixty days after the intervention
  Evaluation of the development of clinical reasoning of nursing students. The instrument Lasater Clinical Judgment Rubric (LCJR) - Brazilian Version will be used. It assesses 11 dimensions at four levels of clinical judgment (recognition, interpretation, response, reflection). The total score ranges from 11 to 44, where the "initial" level generates one point, the "in development" level generates two points, the "proficient" level generates three points and the "exemplary" level generates four points .
Self-efficacy (Baseline) | Applied before the intervention
  Assessment of satisfaction, learning, individual performance after educational actions. A self-efficacy scale will be used. IT'S self-applicable and has 13 items related to beliefs about their own abilities, motivation for action, coping with obstacles, predisposition to challenge, openness to experience, resilience in the face of failures, the influence of initial success on the the final success of an activity and the history of previous successes. These items are represented by a Likert-type scale of agreement, containing five points, in which 1 represents the participant's total disagreement and 5 the total agreement. Scores above 2.5 indicate that participants feel very capable.
Self-efficacy | Applied immediately after the intervention
  Assessment of satisfaction, learning, individual performance after educational actions. A self-efficacy scale will be used. IT'S self-applicable and has 13 items related to beliefs about their own abilities, motivation for action, coping with obstacles, predisposition to challenge, openness to experience, resilience in the face of failures, the influence of initial success on the the final success of an activity and the history of previous successes. These items are represented by a Likert-type scale of agreement, containing five points, in which 1 represents the participant's total disagreement and 5 the total agreement. Scores above 2.5 indicate that participants feel very capable.
Self-efficacy | Applied thirty days after the intervention
  Assessment of satisfaction, learning, individual performance after educational actions. A self-efficacy scale will be used. IT'S self-applicable and has 13 items related to beliefs about their own abilities, motivation for action, coping with obstacles, predisposition to challenge, openness to experience, resilience in the face of failures, the influence of initial success on the the final success of an activity and the history of previous successes. These items are represented by a Likert-type scale of agreement, containing five points, in which 1 represents the participant's total disagreement and 5 the total agreement. Scores above 2.5 indicate that participants feel very capable.
Self-efficacy | Applied sixty days after the intervention
  Assessment of satisfaction, learning, individual performance after educational actions. A self-efficacy scale will be used. IT'S self-applicable and has 13 items related to beliefs about their own abilities, motivation for action, coping with obstacles, predisposition to challenge, openness to experience, resilience in the face of failures, the influence of initial success on the the final success of an activity and the history of previous successes. These items are represented by a Likert-type scale of agreement, containing five points, in which 1 represents the participant's total disagreement and 5 the total agreement. Scores above 2.5 indicate that participants feel very capable.

SECONDARY OUTCOMES:
Student stress (Baseline) | Before the intervention
  Assessment of the intensity of stress among nursing students caused by pedagogical strategies: high-fidelity simulation and digital educational platforms. The questionnaire will be applied. It consists of 31 items and the answers are Likert type, scored from 0 to 3, depending on the degree of concern it generates for the student, as follows: nothing (0), a little (1), a lot (2) and extremely ( 3).
Student stress | Applied immediately after the intervention
  Assessment of the intensity of stress among nursing students caused by pedagogical strategies: high-fidelity simulation and digital educational platforms. The questionnaire will be applied. It consists of 31 items and the answers are Likert type, scored from 0 to 3, depending on the degree of concern it generates for the student, as follows: nothing (0), a little (1), a lot (2) and extremely ( 3).
Student stress | Applied thirty days after the intervention
  Assessment of the intensity of stress among nursing students caused by pedagogical strategies: high-fidelity simulation and digital educational platforms. The questionnaire will be applied. It consists of 31 items and the answers are Likert type, scored from 0 to 3, depending on the degree of concern it generates for the student, as follows: nothing (0), a little (1), a lot (2) and extremely ( 3).
Student stress | Applied sixty days after the intervention
  Assessment of the intensity of stress among nursing students caused by pedagogical strategies: high-fidelity simulation and digital educational platforms. The questionnaire will be applied. It consists of 31 items and the answers are Likert type, scored from 0 to 3, depending on the degree of concern it generates for the student, as follows: nothing (0), a little (1), a lot (2) and extremely ( 3).

CONTACTS AND LOCATIONS:
Overall Officials: Marcia CS Magro, PhD, Principal Investigator — University of Brasilia

REFERENCES:
- [Background] Silveira MS, Cogo ALP. The contributions of digital technologies in the teaching of nursing skills: an integrative review. Rev Gaucha Enferm. 2017 Jul 13;38(2):e66204. doi: 10.1590/1983-1447.2017.02.66204. English, Portuguese. PMID 28723986
- [Background] Basak T, Unver V, Moss J, Watts P, Gaioso V. Beginning and advanced students' perceptions of the use of low- and high-fidelity mannequins in nursing simulation. Nurse Educ Today. 2016 Jan;36:37-43. doi: 10.1016/j.nedt.2015.07.020. Epub 2015 Jul 29. PMID 26282193
- [Background] Cogo ALP, Lopes EFDS, Perdomini FRI, Flores GE, Santos MRRD. Building and developing realistic simulation scenarios on safe drug administration. Rev Gaucha Enferm. 2019 Jan 10;40(spe):e20180175. doi: 10.1590/1983-1447.2019.20180175. English, Portuguese. PMID 30652802
- [Background] Valentin B, Grottke O, Skorning M, Bergrath S, Fischermann H, Rortgen D, Mennig MT, Fitzner C, Muller MP, Kirschbaum C, Rossaint R, Beckers SK. Cortisol and alpha-amylase as stress response indicators during pre-hospital emergency medicine training with repetitive high-fidelity simulation and scenarios with standardized patients. Scand J Trauma Resusc Emerg Med. 2015 Apr 8;23:31. doi: 10.1186/s13049-015-0110-6. PMID 25887044
- [Background] McGuire K, Lorenz R. Effect of Simulation on Learner Stress as Measured by Cortisol: An Integrative Review. Nurse Educ. 2018 Jan/Feb;43(1):45-49. doi: 10.1097/NNE.0000000000000393. PMID 28538244
- [Background] Fraser K, McLaughlin K. Temporal pattern of emotions and cognitive load during simulation training and debriefing. Med Teach. 2019 Feb;41(2):184-189. doi: 10.1080/0142159X.2018.1459531. Epub 2018 Apr 24. PMID 29687734
- [Background] Nieto Fernandez-Pacheco A, Castro Delgado R, Arcos Gonzalez P, Navarro Fernandez JL, Ceron Madrigal JJ, Juguera Rodriguez L, Perez Alonso N, Armero-Barranco D, Lidon Lopez Iborra M, Damian ET, Pardo Rios M. Analysis of performance and stress caused by a simulation of a mass casualty incident. Nurse Educ Today. 2018 Mar;62:52-57. doi: 10.1016/j.nedt.2017.12.016. Epub 2017 Dec 15. PMID 29291462
- [Background] Mohammadi G, Tourdeh M, Ebrahimian A. Effect of simulation-based training method on the psychological health promotion in operating room students during the educational internship. J Educ Health Promot. 2019 Sep 30;8:172. doi: 10.4103/jehp.jehp_106_19. eCollection 2019. PMID 31867357
- [Background] de Sena DP, Fabricio DD, da Silva VD, Bodanese LC, Franco AR. Comparative evaluation of video-based on-line course versus serious game for training medical students in cardiopulmonary resuscitation: A randomised trial. PLoS One. 2019 Apr 8;14(4):e0214722. doi: 10.1371/journal.pone.0214722. eCollection 2019. PMID 30958836
- [Background] Blanie A, Amorim MA, Meffert A, Perrot C, Dondelli L, Benhamou D. Assessing validity evidence for a serious game dedicated to patient clinical deterioration and communication. Adv Simul (Lond). 2020 May 27;5:4. doi: 10.1186/s41077-020-00123-3. eCollection 2020. PMID 32514382
- [Background] Fonseca LM, Aredes ND, Fernandes AM, Batalha LM, Apostolo JM, Martins JC, Rodrigues MA. Computer and laboratory simulation in the teaching of neonatal nursing: innovation and impact on learning. Rev Lat Am Enfermagem. 2016 Oct 10;24:e2808. doi: 10.1590/1518-8345.1005.2808. PMID 27737376